CLINICAL TRIAL: NCT01225250
Title: An Open-Label, Randomized, 2-Arm Parallel Study Comparing the Efficacy, Ease of Use, and Safety of PDS Plated Cartilagenous Grafting Versus Non-Plated Cartilagenous Grafting as Performed Through Endonasal Rhinoplasty
Brief Title: Safety and Efficacy Study of Polydioxanone (PDS) Plates in Rhinoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Principal Investigator, Steven H. Dayan, Medical Director, DeNova Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDS-END-001
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Rhinoplasty
Keywords: Caudal septal extension graft; Primary rhinoplasty; Secondary rhinoplasty
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polydioxanone (PDS) plates (Experimental): 15 subjects will be randomized to receive a caudal septal extension graft using a PDS plated cartilagenous graft
  Interventions: Device: Polydioxanone (PDS) plates; Procedure: Caudal septal extension graft performed through endonasal rhinoplasty
- Non-plated cartilagenous graft (Other): 15 subjects will be randomized to receive a cartilagenous caudal septal extension fgraft
  Interventions: Procedure: Caudal septal extension graft performed through endonasal rhinoplasty

INTERVENTIONS:
Device: Polydioxanone (PDS) plates — 0.5 mm PDS Flexible Plate made of poly-p-dioxanone, an aliphatic polyester which is manufactured by polymerization of the monomer p-dioxanone. Polydioxanone is a resorbable material degraded by hydrolysis and has been successfully used for bone discontinuities and septal reconstruction.
  Arms: Polydioxanone (PDS) plates
Procedure: Caudal septal extension graft performed through endonasal rhinoplasty — The caudal septal extension (CSE) graft is a common method used to alter tip projection, alar-columellar relationship, and nasolabial angle.5 However, it can be difficult to stabilize and straighten the CSE graft, especially when performed through an endonasal approach. Use of a polydioxanone plate would provide a scaffolding for the CSE graft and could allow for a technically easier and more predictable surgical procedure.
  Arms: Polydioxanone (PDS) plates
Procedure: Caudal septal extension graft performed through endonasal rhinoplasty — The caudal septal extension (CSE) graft is a common method used to alter tip projection, alar-columellar relationship, and nasolabial angle.5 However, it can be difficult to stabilize and straighten the CSE graft, especially when performed through an endonasal approach. Use of a polydioxanone plate would provide a scaffolding for the CSE graft and could allow for a technically easier and more predictable surgical procedure.
  Arms: Non-plated cartilagenous graft

SUMMARY:
The purpose of this study is to determine efficacy, safety, and ease of cartilaginous grafting using polydioxanone (PDS) plates in comparison to non-plated cartilaginous grafts as performed through an endonasal rhinoplasty approach in patients requiring a caudal septal extension (CSE) graft.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age.
* Subjects requesting primary or secondary rhinoplasty and requiring a CSE graft performed through an endonasal approach.
* Subjects willing to undergo PDS plating.
* Subjects with either ear conchal or septal cartilage available for grafting purposes.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Willingness and ability to comply with the PI's standard preoperative and postoperative rhinoplasty instructions.
* Subjects of childbearing potential must have a negative urine pregnancy test result at Visit 1 and be willing able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following is documented on the medical history:
* postmenopausal for at least 12 months prior to study drug administration
* without a uterus and/or both ovaries
* has had a bilateral tubal ligation for at least 6 months prior to study drug administration.
* absence of an other physical condition according to the PI's discretion
* Willingness and ability to provide written photo consent and adherence to photography procedures (i.e., removal of jewelry and makeup).
* Willingness and ability to provide written informed consent prior to performance of any study related procedure.

Exclusion Criteria:

* Subjects who are pregnant, nursing, planning to become pregnant, and/or not using a reliable form of birth control.
* Subjects with a significant systemic illness or illness localized to the areas of treatment.
* Subjects with previous history of nasal implants.
* Subjects with previous or current history of nasal infections.
* Subjects who have history of blood thinners (aspirin, ibuprofen, naprosyn, herbal supplements, Vitamin E) within the two weeks prior to surgery.
* Subjects who have smoked within the two weeks prior to surgery.
* Subjects who have had alcohol or illicit drugs one week prior to surgery.
* Subjects who have eaten or drank anything after midnight the night prior to surgery.
* Subjects with current history of chronic drug or alcohol abuse.
* History of autoimmune disease.
* Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study medication.
* Subjects who anticipate the need for surgery, other than the study procedure, or overnight hospitalization during the study.
* Subjects who, in the Investigator's opinion, have a history of poor cooperation, non compliance with medical treatment or unreliability.
* Enrollment in any active study involving the use of investigational devices or drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-11-24 (Actual); Primary Completion 2015-01-19 (Actual); Study Completion 2015-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Dayan, MD, Principal Investigator — DeNova Research/ Chicago Center for Facial Plastic Surgery
Locations (1):
- DeNova Research, Chicago, Illinois, United States

REFERENCES:
- [Derived] Dayan SH, Ashourian N. Polydioxanone Absorbable Plate for Cartilaginous Grafting in Endonasal Rhinoplasty: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2016 Jan-Feb;18(1):47-53. doi: 10.1001/jamafacial.2015.1492. PMID 26501937
- See also: DeNova Research — http://www.denovaresearch.com
- See also: Dr. Steven H. Dayan, MD FACS — http://www.drdayan.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Started | 15 | 15
Completed | 10 | 10
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 49 [23 to 64] | 48 [29 to 62] | 48.5 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Live Assessment of Satisfaction With the Grafts
Description: Efficacy will be determined by a live assessment of satisfaction with the grafts at 12 months using a four-point categorical satisfaction scale ((4) unsatisfied, (3) satisfied, (2) very satisfied, (1) highly satisfied).
  Scores closer to 1 indicate a more favorable outcome
Time Frame: 12 months post operative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
units on a scale | 2 (0.667) | 4 (0.05)

2. Primary Outcome: Assessment of Tip Projection
Description: Tip projection will be measured using standardized photography preoperatively and at 1 month, 3 months, 6 months, and 12 months postoperatively using Goode's Ratio.
  The ratio of the line from the alar crease to the nasal tip to the nasion to the nasal tip should be 0.55. If it is more than that the nose is over projected, if it is under that ratio the nose is under projected.
Time Frame: 12 months Post opeartive
Measure: Mean (Standard Deviation); unit: ratio of tip projection to nasal length
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
ratio of tip projection to nasal length
  Month 1 | 0.55 (0.6) | 0.58 (0.05)
  Month 3 | 0.54 (0.06) | 0.58 (0.04)
  Month 6 | 0.54 (0.05) | 0.57 (0.03)
  Month 12 | 0.55 (0.06) | 0.55 (0.05)

3. Primary Outcome: Non-treating Blinded Evaluator Satisfaction Assessment
Description: A non-treating blinded evaluator will assess satisfaction with a four-point categorical satisfaction scale ((4) - unsatisfied, (3) - satisfied, (2) - very satisfied, (1) - highly satisfied) of subject's grafts using photographs from baseline, 1 month, 3 months, 6 months, and 12 months and will consist of a blinded evaluation in which the physician is aware of the type of graft, but unaware of plating status or the specific grafting site.
  Scores closer to 1 indicate a more favorable outcome
Time Frame: Assessed at baseline, 1 month, 3 months, 6 months, and 12 months; Month 12 reported
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
score on a scale | 2 (1) | 2 (1)

4. Primary Outcome: Ease of Use
Description: Ease of use will be determined by the treating investigator using a 10 cm Visual Analog Scale (VAS) to demonstrate technical ease with a score of 0 mm being easy and a scale of 100 mm being extremely difficult.
Time Frame: 1 hour following surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
score on a scale | 17 (9.95) | 46.4 (13.43)

5. Secondary Outcome: Number of Participants With Infection, Rejection, and Extrusion of the Graft at 1 Week, 1 Month, 3 Months, 6 Months, and 12 Months
Description: Safety will be determined by rate of infection, rejection, and extrusion of the graft at 1 week, 1 month, 3 months, 6 months, and 12 months.
Time Frame: 12 months post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
Participants
  Week 1 - Infection | 0 | 1
  Week 1 - Rejection | 0 | 0
  Week 1 - Extrusion | 0 | 0
  Month 1 - Infection | 1 | 0
  Month 1 - Rejection | 0 | 0
  Month 1 - Extrusion | 0 | 0
  Month 3 - Infection | 0 | 0
  Month 3 - Rejection | 0 | 0
  Month 3 - Extrusion | 0 | 0
  Month 6 - Infection | 0 | 0
  Month 6 - Rejection | 0 | 0
  Month 6 - Extrusion | 0 | 0
  Month 12 - Infection | 0 | 0
  Month 12 - Rejection | 0 | 0
  Month 12 - Extrusion | 0 | 0

6. Secondary Outcome: Intraoperative Duration
Description: The intraoperative duration of the grafting procedure will be measured by an assistant using a stopwatch to record the time it takes to harvest, shape, and satisfactorily secure the graft.
Time Frame: During surgery (up to 3 hours)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
Number analyzed (Participants) | 15 | 15
seconds | 604.7 (219.12) | 571.5 (182.16)

ADVERSE EVENTS:
Arm/Group | Polydioxanone (PDS) Plates | Non-plated Cartilagenous Graft
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes